CLINICAL TRIAL: NCT07079241
Title: REgion Skåne Preventing Overdose Through Naloxone Distribution With Emergency Runners: a Feasibility Study for a Model to Save Lives Through a Volunteer First Responder Service Providing Antidote Treatment in Opioid Overdose
Brief Title: A Model to Save Lives Through a Volunteer First Responder Service Providing Antidote Treatment in Opioid Overdose
Acronym: RESPONDER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: SOS Alarm Sverige AB (Unknown); Lund University (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-05887-01
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-06

CONDITIONS: Opioid Overdose
Keywords: Opioid overdose; Community first responder; Volunteer first responder; Medical emergency; Dispatcher; Naloxone; Overdose; Intoxication; Smartphone applications; First responder system; Emergency medical dispatcher
MeSH Terms: conditions — Opiate Overdose; Drug Overdose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Naloxone-responders (Experimental): Naloxone-responder is the name of a volunteer first responder who participate in the study. These participants will fulfill a pre-registration course on overdose and opioid recognition, naloxone usage and first aid education following European and national guidelines. The participants will also be educated in low-arousal approaches to beneficially meet and communicate with potential overdose victims. Naloxone-responders will be equipped with a kit containing two doses of nasal naloxone and registered as active users on the unique RESPONDER application. Minimum age is 18 years old to become a responder.
  Interventions: Other: Naloxone-responder: A volunteer first responder system connected to emergency dispatch service and alerting overdose and first aid educated volunteers with naloxone to suspected opioid overdoses

INTERVENTIONS:
Other: Naloxone-responder: A volunteer first responder system connected to emergency dispatch service and alerting overdose and first aid educated volunteers with naloxone to suspected opioid overdoses — The model is a smartphone-based alert system with an app which is connected to dispatcher centers. Volunteer first responders will be alerted in addition to standard emergency medical service (like ambulance) to suspected opioid overdoses and also cardiac arrests. The aim is to see if volunteers equipped with naloxone and with up-do-date knowledge of overdose treatment and first aid can arrive and reverse the condition safely prior to emergency service arrival.

SUMMARY:
Opioids are responsible for the greatest drug-related global health burden. Prevention and treatment programs for people with opioid use disorder are widely implemented, but further actions are required to reduce the mortality and morbidity caused by opioid use and dependence. We suggest a novel and unique approach with a volunteer first responder system for suspected opioid overdoses, integrated with national emergency call services. The idea derives from the success of volunteer first responder systems for out-of-hospital cardiac arrests. Several reports exist globally with results of increased survival rates, less complications and a beneficial time-gain to start of cardiopulmonary resuscitation before emergency services (like ambulance and fire fighters) arrival.

Our model aims to investigate feasibility, acceptability and safety of a smartphone-based volunteer first responder system for suspected opioid overdoses. The volunteer responders will be equipped with an emergency kit including two doses of the opioid antidote naloxone, which can reverse life-threatening respiratory arrest caused by intoxication of opioids. The responders will, prior to registration, accomplish an in-depth overdose and naloxone education, as well as a first aid course aligned with current European and Swedish resuscitation guidelines. The results will be collected through questionnaires to the responder participants, technical data from the responder application, and dispatcher, pre-medical/paramedical and hospital records among others. Both quantitative and qualitative methods will be used. The major question is if the model is feasible in alerting lay persons with naloxone to suspected overdose situations and successfully administer naloxone prior to emergency service arrival. Furthermore, experiences of safety during alerts among volunteer first responders and overdose victims will also be studied.

Our model is unique in its integration with emergency medical dispatch service along with overdose and first aid education prior to participant registration. The respiratory arrest of opioids is an acute life-threatening condition, which - in similarity to cardiac arrests - need emergent actions for survival. A reduced time to naloxone administration through volunteer first responders prior to ambulance arrival could save lives.

DETAILED DESCRIPTION:
The accuracy of opioid overdose recognition among medical dispatchers is as of today an underexplored field. The risk of naloxone-responders being alerted to other medical emergencies than opioid overdoses is as a consequence unknown. The first aid course aims to improve the knowledge and emergency management of responders who get alerted to false positive opioid overdoses, while the naloxone and overdose in-depth education aims to help responders to properly identify and manage true overdoses.

Naloxone reverses opioid effects temporally, which calls for prolonged medical assistance with observation and sometimes repeated doses of naloxone at the hospital. The integration of naloxone-responder alerts and emergency medical service dispatching when bystander call the national emergency number is therefore a model with both short- and long-term management of overdose conditions.

The RESPONDER trial is a two-year pilot project with a one-year follow-up of each registered participant, so called naloxone-responder. At least four different follow-up sub-studies will be performed during and 1-2 years after the pilot period:

1. A quantitative study of feasibility, acceptability and safety of the intervention.
2. A quantitative study on mortality post-pilot as primary outcome, and clinical outcome after intervention compared to no intervention as secondary outcome.

3 and 4. Two qualitative studies exploring the experiences of: A. receiving naloxone from a naloxone-responder, from the overdose survivors' point of view, and B. accepting overdose alerts as a naloxone-responder, respectively.

ELIGIBILITY:
Inclusion Criteria for volunteer first responder:

1. Give informed written consent to participate in the study
2. Successfully complete an opioid overdose and naloxone course in addition to a first aid course, following current first aid guidelines from the Swedish Resuscitation Council and the European Resuscitation Council.
3. Download and register oneself as a user on the project-specific volunteer first responder app on a smartphone
4. Purchase naloxone from a pharmacy and receive reimbursement for the full cost of the purchase upon submission of the pharmacy receipt

Exclusion Criteria for volunteer first responder:

1. Displaying inappropriate behavior during the education day (or otherwise in time, as witnessed or experienced by course instructors or the project team). Such conduct could for example be to not follow the guidelines of low-arousal (non-confrontational) approach in emergencies.

Inclusion Criteria for overdose alerts:

1. Victim being ≥15 years old
2. Any naloxone-responder being up to 10.000 meters from the situation, in Skåne

Exclusion Criteria for overdose alerts:

1. Any trauma behind the condition
2. Dispatcher impression of the scene to be unsafe for lay persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of successful naloxone-responder alerts to true opioid overdoses | 12 months of participation for every registered naloxone-responder
  Emergency calls with dispatchers' activation of alerts to naloxone-responders who manage to administer naloxone in situations of true opioid overdoses prior to EMS arrival
Positioning of and acceptability of alerts among naloxone-responders equipped with naloxone in relation to overdose locations | Data during 12 months from registration for every naloxone-responder
  Distance between naloxone-responders and emergency scenes when receiving alerts and the frequency of accepting or rejecting the notification among responders with versus without their naloxone-kit on hand
Clinical outcome of overdose victims before versus after the trial | Data compared 1.5-2 years post trial start.
  Mental and clinical status, morbidity and survival rates from questionaires and medical records during the trial, compared to historic control period.
Safety and acceptability as experienced by naloxone-responders and overdose victims | Ongoing during the trial period of one year for every naloxone-responder and overdose victim during the time. A second survey 12-months post-registration for every naloxone-responder.
  Experience of being at the scene from two different perspectives, with views collected through questionaires post-alerts and qualitative interviews post-trial.

SECONDARY OUTCOMES:
Mortality rates before versus after the trial | 1-2 years from trial start, compared to 1-3 years prior to trial start.
  Current regional statistics post-trial and pre-trial.

CONTACTS AND LOCATIONS:
Overall Officials: Anders C Håkansson, MD, prof., Principal Investigator — Malmö Addiction Center, Region Skåne, Sweden
Locations (1):
- Malmö Addiction Center, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No